CLINICAL TRIAL: NCT06648694
Title: Correlation Between Intra-abdominal Pressure and Diaphragmatic Mobility in Women Submitted to Abdominoplasty After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Sandra Fluhr Souto Barros, PhD Student, Universidade Federal de Pernambuco
Other Study IDs: UFPernambucoCirDoutorado
Record Dates: First submitted 2023-12-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Abdominoplasty Surgery
Keywords: Abdominoplasty; Abdominal Dermolipectomy; Bariatric Surgery; Obesity; Diaphragmatic Mobility; Intra-abdominal Pressure
MeSH Terms: conditions — Obesity | interventions — Abdominoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Abdominoplasty surgery — Correlation between IAP and Diaphragmatic Mobility
Procedure: Abdominoplasty — For the practice of the surgical procedure, the region to be operated on was marked using a surgical marking pen (Textel®). With the patient in the orthostatic position, a median line was drawn from the xiphoid appendix to the pubic symphysis, reaching the anterior vulvar commissure. Then, with the patient in the dorsal position, a transverse line was drawn 6 cm above the vulvar commissure and elongated to the iliac spine on each side. From there, the lateral skin surplus was estimated by means of bidigital clamping. The excess tissue was marked in a triangular shape, with a slight arching up to the xiphoid appendix. To determine the horizontal skin surplus, marking was performed, similar to that performed in classic abdominoplasty described in the literature(AMORIM FILHO; AMORIM, 2012). In this study, an anchor incision was recommended for all volunteers. All patients underwent intravenous sedation followed by spinal anesthesia.

SUMMARY:
Background: Plication of the rectus abdominis muscles leads to an increase in intra-abdominal pressure (IAP), which may negatively impact the respiratory system due to its effects on diaphragmatic mobility (DM).

Objective: To establish the correlation between IAP following plication of the rectus abdominis muscles and DM in women who have undergone abdominoplasty after bariatric surgery.

Methods: This prospective cohort study evaluated DM and IAP using high-resolution ultrasound and intravesical pressure measurement during the preoperative, intraoperative, and 1st postoperative day (POD1) periods. Hypotheses: There is a negative correlation between intra-abdominal pressure values after plication of the rectus abdominis muscles and diaphragmatic mobility. There is an increase in intra-abdominal pressure after plication of the rectus abdominis muscles, which is aggravated by the modified Fowler position and the use of the compression belt. The greater the width of the diastasis, the greater the IAP.

DETAILED DESCRIPTION:
Introduction:

Plication of the rectus abdominis muscles leads to an increase in intra-abdominal pressure (IAP), which may negatively impact the respiratory system due to its effects on diaphragmatic mobility (DM).

Objective: To establish the correlation between IAP following plication of the rectus abdominis muscles and DM in women who have undergone abdominoplasty after bariatric surgery.

hypotheses:

The present study has the following hypotheses:

I. There is a negative correlation between intra-abdominal pressure values after plication of the rectus abdominis muscles and diaphragmatic mobility.

II. There is an increase in intra-abdominal pressure after plication of the rectus abdominis muscles.

III. The increase in intra-abdominal pressure is aggravated by the modified Fowler positioning.

IV. There is a positive correlation between diastasis width and intra-abdominal pressure.

V. Diaphragmatic mobility in the immediate postoperative period is reduced when compared to the preoperative period.

VI. The use of the compression belt increases intra-abdominal pressure. VII. There is a positive correlation between intra-abdominal pressure values and pain.

Objective: To establish the correlation between IAP following plication of the rectus abdominis muscles and DM in women who have undergone abdominoplasty after bariatric surgery.

Methods:

This is a prospective cohort study conducted in the surgical center of Hospital Agamenon Magalhães (HAM) in partnership with its plastic surgery outpatient clinic, from August 2017 to March 2020. The study evaluated intra-abdominal pressure in the preoperative period, immediately after plication of the rectus abdominis muscles in the supine position, post-plication of the rectus abdominis muscles in a modified Fowler's position, post-plication of the rectus abdominis muscles after complete abdominal suturing, post-abdominal bandaging, and on the 1st postoperative day (POD) with and without a compression garment, in healthy women undergoing abdominoplasty after gastroplasty.

This project was approved by the Research Ethics Committee of the Health Sciences Center at HC-UFPE (CAAE: 68563416.5.3001.5197). All participants included in this study met the eligibility criteria and signed the informed consent form.

The study included women aged 25 to 55 years old who underwent abdominoplasty after bariatric surgery under spinal anesthesia, with an anchor-shaped scar, presenting type IV or V abdominal deformity as described by Bozola [23], with stable body weight for a minimum of 6 months after achieving post-bariatric surgery weight loss goals, and a body mass index (BMI) ≤ 30 kg/m2. All study participants scored above 18 points on the Mini-Mental State Examination. Patients with respiratory and cardiac comorbidities and a history of smoking for more than 10 years were excluded from the analysis.

The primary outcomes analyzed were intra-abdominal pressure (IAP), expressed in millimeters of mercury (mmHg), and diaphragmatic mobility (DM), expressed in millimeters (mm). Secondary outcomes included the evaluation of dyspnea and pain levels.

Intra-abdominal pressure was measured during the preoperative period, immediately after plication of the rectus abdominis muscles with the abdomen open in the supine position and then in a modified Fowler's position, after abdominal wall synthesis, after bandaging, and on the 1st postoperative day with and without a compression garment. Diaphragmatic mobility, pain intensity, and dyspnea were evaluated in the preoperative period and on the 1st postoperative day.

Initially, anamnesis and physical examination were performed on all volunteers during the preoperative period, where personal data and anthropometric measurements were recorded: weight (Kg), height (m), and BMI; and vital signs: Respiratory Rate (RR) (rpm), Heart Rate (HR) (Bpm), Blood Pressure (BP) (mmHg), and Peripheral Oxygen Saturation (SPO2).

Since intravesical pressure measurement reflects intra-abdominal pressure, we measured it at the intraoperative periods mentioned earlier and on the 1st postoperative day. After obtaining bladder catheterization using a 16 Fr 3-way Foley catheter (Sisco®) with the outflow channel properly clamped, we connected the intermediate channel to a device composed of an intravenous infusion set (Hartmann®), which was attached to a calibrated stand with the zero mark positioned at the level of the patient's pubic symphysis.

This set was connected to a 0.9% sodium chloride solution bag for the injection of 50 ml of saline solution after bladder emptying at each measurement stage.

Thus, IAP was measured in cmH2O 30 seconds after saline infusion to obtain the pressure measurement after detrusor muscle relaxation of the bladder. This pressure was later converted to mmHg (1 cmH2O = 0.74 mmHg).

To assess diaphragmatic mobility, a high-resolution ultrasound device (Philips - HD11 XE) with a 3.5 MHz convex transducer was used, following the protocol described by Testa et al. The volunteers then received verbal instructions to perform forced vital capacity maneuvers, where the measurement of each curve, corresponding to the displacement of the diaphragmatic blade, was performed immediately after obtaining the images. The maneuvers were repeated until 5 satisfactory images were obtained. A mean of the 3 highest values was used, provided that these did not differ by more than 10% from each other. All DM measurements were performed by the same evaluator.

The Visual Analog Scale (VAS) was used to assess postoperative pain intensity. Patients were asked about their perception of dyspnea through the Modified Borg Scale, following the recommendations of the American Thoracic Society.

ELIGIBILITY:
The study included women aged 25 to 55 years old who underwent abdominoplasty after bariatric surgery under spinal anesthesia, with an anchor-shaped scar, presenting type IV or V abdominal deformity as described by Bozola, with stable body weight for a minimum of 6 months after achieving post-bariatric surgery weight loss goals, and a body mass index (BMI) ≤ 30 kg/m2. All study participants scored above 18 points on the Mini-Mental State Examination. Patients with respiratory and cardiac comorbidities and a history of smoking for more than 10 years were excluded from the analysis.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing abdominal dermolipectomy surgery after gastroplasty who meet the eligibility criteria for the search.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic Mobility | preoperative and on the 1st postoperative day.
  Measure diaphragmatic mobility for total lung capacity maneuver
Intraabdominal Pressure | preoperatively, after plication of the rectus abdominis muscles in the supine and modified Fowler positions, after abdominal wall synthesis, after bandaging and on the 1st postoperative day with and without girdle.
  evaluated intra-abdominal pressure in the preoperative period, immediately after plication of the rectus abdominis muscles in the supine position, post-plication of the rectus abdominis muscles in a modified Fowler's position, post-plication of the rectus abdominis muscles after complete abdominal suturing, post-abdominal bandaging, and on the 1st postoperative day (POD) with and without a compression garment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sandra Fluhr, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No